CLINICAL TRIAL: NCT06284720
Title: Transcranial Alternating Current Stimulation for the Improvement of Episodic Memory in Healthy Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica Portuguesa (Other)
Collaborators: Clínica NeuroVida (Portugal) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Project number 144
Record Dates: First submitted 2024-01-27; First posted 2024-02-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy Older Adults
Keywords: healthy aging; episodic memory; gamma oscillations; transcranial alternating current stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: real tACS (Experimental): 5 sessions of gamma tACS (40 Hz) at 2 mA over the Precuneus
  Interventions: Device: Gamma tACS (40 Hz) over the precuneus
- Placebo Comparator: sham tACS (Sham Comparator): 5 sessions of sham over the Precuneus
  Interventions: Device: Sham tACS over the precuneus

INTERVENTIONS:
Device: Gamma tACS (40 Hz) over the precuneus — 5 sessions of gamma tACS (40 Hz) over the precuneus
  Arms: Experimental: real tACS
Device: Sham tACS over the precuneus — 5 sessions of sham tACS over the precuneus
  Arms: Placebo Comparator: sham tACS

SUMMARY:
Memory complaints are a common symptom among Subjective Cognitive Decline, Mild Cognitive Impairment and Alzheimer disease. Indeed, episodic memory and Alzheimer disease are highly sensitive to aging. Many brain areas become active when we remember an event from the past. The precuneus, part of the posterior system of default mode network, has been identified as a central node of episodic memory retrieval and a central node in various psychiatric and neurological disorders, such as Alzheimer disease. Age-related changes have been consistently found in the default mode network connectivity, occurring within its posterior areas and with the reduction of connectivity between anterior and posterior subnetwork. It has also been found that aging is associated with decreased functional connectivity in the precuneus and posterior cingulate of the default mode network. Furthermore, γ-Aminobutyric acid (GABA), which plays an essential role in regulating brain activity and modulating the default mode network, shows a decrease throughout the normal course of aging, in Mild Cognitive Impairment and Alzheimer disease. It was also verified a link between cognitive decline and the dysfunction of the inhibitory activity of GABAergic interneurons, particularly parvalbumin-positive interneurons, that play a role in control local circuitry, brain networks and memory processing. Parvalbumin interneurons are the fast-spiking interneurons that generate and maintain gamma frequency. Gamma band has been associated with the encoding and retrieval of episodic memory. Impairments of gamma oscillations have been observed in healthy aging, Mild Cognitive Impairment and Alzheimer disease.

By identifying these functional connectivity changes, non-invasive neuromodulation techniques may offer a new strategy for improving cognitive functions. Transcranial Alternating Current Stimulation (tACS) is a form of non-invasive brain stimulation that modulates cortical activity by applying weak, oscillating electrical currents to the cortex via two or more scalp electrodes. By using alternating currents, it is possible to simulate the rhythmic pattern of electrophysiological activity of the brain. tACS can interact with neural firing at behaviorally relevant frequencies linked to memory.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate whether stimulation with gamma tACS on the precuneus can improve episodic memory in healthy older adults.

DETAILED DESCRIPTION:
Memory complaints are a common symptom among Subjective Cognitive Decline, Mild Cognitive Impairment and Alzheimer disease. Indeed, episodic memory and Alzheimer disease are highly sensitive to aging. Many brain areas become active when we remember an event from the past. The precuneus, part of the posterior system of default mode network, has been identified as a central node of episodic memory retrieval and a central node in various psychiatric and neurological disorders, such as Alzheimer disease. Age-related changes have been consistently found in the default mode network connectivity, occurring within its posterior areas and with the reduction of connectivity between anterior and posterior subnetwork. It has also been found that aging is associated with decreased functional connectivity in the precuneus and posterior cingulate of the default mode network. Furthermore, γ-Aminobutyric acid (GABA), which plays an essential role in regulating brain activity and modulating the default mode network, shows a decrease throughout the normal course of aging, in Mild Cognitive Impairment and Alzheimer disease. It was also verified a link between cognitive decline and the dysfunction of the inhibitory activity of GABAergic interneurons, particularly parvalbumin-positive interneurons, that play a role in control local circuitry, brain networks and memory processing. Parvalbumin interneurons are the fast-spiking interneurons that generate and maintain gamma frequency. Gamma band has been associated with the encoding and retrieval of episodic memory. Impairments of gamma oscillations have been observed in healthy aging, Mild Cognitive Impairment and Alzheimer disease.

By identifying these functional connectivity changes, non-invasive neuromodulation techniques may offer a new strategy for improving cognitive functions. Transcranial Alternating Current Stimulation (tACS) is a form of non-invasive brain stimulation that modulates cortical activity by applying weak, oscillating electrical currents to the cortex via two or more scalp electrodes. By using alternating currents, it is possible to simulate the rhythmic pattern of electrophysiological activity of the brain. tACS can interact with neural firing at behaviorally relevant frequencies linked to memory.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate whether stimulation with gamma tACS on the precuneus can improve episodic memory in healthy older adults.

Participants will be randomized into two groups in a 1:1 ratio, and the order of administration of either intervention (i.e., gamma-tACS or sham) will be counterbalanced across all participants. Stimulation will be inverted (crossover phase) after 1 week (wash-out). Participants will be evaluated with neuropsychological tests (AVLT and FNMT) and neurophysiological measures of functional connectivity (rs EEG).

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 or over;
* Normal general cognition: score within the normative values for the Portuguese population in the Addenbrooke's Cognitive Examination

Exclusion Criteria:

* Neurological disorders (stroke, tumours, significant head trauma, and epilepsy), psychiatric conditions (such as autism, schizophrenia, depression), or uncontrolled medical illness (hypertension, metabolic, endocrine, toxic, and infectious diseases) able to interfere with cognition;
* Sensory deficits likely to interfere with neuropsychological assessment;
* Impairment in activities of daily living;
* Chronic alcohol or drug abuse;
* Non-native Portuguese speakers;
* Metal implants on the head or implanted electronic devices.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in immediate and delayed free recall Auditory Verbal Learning Test scores | Baseline (immediately before the stimulation protocol/on the first session/day 1) and post stimulation (after 5 sessions of 5 consecutive days of gamma tACS/sham/day 5). After one week, measures will be repeated in the crossover phase day 12 and 17.
  Auditory Verbal Learning Test is a list-learning paradigm, and consists of five consecutive immediate free recall trials, a delayed free recall trial (after 30 minutes of the fifth immediate free recall trial), and a delayed recognition trial. Different lists will be used during pre- and post-stimulation to avoid learning effects.
Changes in immediate free recall and delayed recognition Face-Name Memory Test scores | During the first session/day 1 of intervention of gamma tACS/sham and during the first session on the crossover-phase/day12
  Face-Name Memory Test requires learning 20 unfamiliar face-name pairs and include a training, initial learning phase (learning 1 and 2), immediate recall and after 30 minutes a delayed recall, facial recognition, and a multiple-choice recognition trial. During learning phase (1 and 2) participants will underwent two exposures to all 20 face and name. It is shown a face on a grey background with a fictional first name printed in black underneath the face, forming a face-name pair; the participants must say whether the photograph they see is of a man or a woman, read the name below out loud and try to learn each face-name pair. Following each exposure, they were asked for name associated with each face. After a 30-minute delay they were asked to identify the previously learned face from three pictures, asked for name associated with each face, and asked to select the name associated with the face among four proper names

SECONDARY OUTCOMES:
Change in functional connectivity | Baseline (immediately before the stimulation protocol/on the first session/day 1) and post stimulation (after 5 sessions of 5 consecutive days of gamma tACS/sham/day 5). After one week, measures will be repeated in the crossover phase day 12 and 17.
  By using resting state electroencephalogram the investigators will evaluate the effects of gamma tACS in functional connectivity between precuneus and hippocampus

CONTACTS AND LOCATIONS:
Locations (1):
- Filipa Ribeiro, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All data, including outcome measure results, study protocol and statistical analysis plan, will be shared upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the study completion indefinitely.
Access Criteria: Reasonable request

REFERENCES:
- [Background] Bai X, Edden RA, Gao F, Wang G, Wu L, Zhao B, Wang M, Chan Q, Chen W, Barker PB. Decreased gamma-aminobutyric acid levels in the parietal region of patients with Alzheimer's disease. J Magn Reson Imaging. 2015 May;41(5):1326-31. doi: 10.1002/jmri.24665. Epub 2014 May 27. PMID 24863149
- [Background] Billette OV, Ziegler G, Aruci M, Schutze H, Kizilirmak JM, Richter A, Altenstein S, Bartels C, Brosseron F, Cardenas-Blanco A, Dahmen P, Dechent P, Dobisch L, Fliessbach K, Freiesleben SD, Glanz W, Goerss D, Haynes JD, Heneka MT, Kilimann I, Kimmich O, Kleineidam L, Laske C, Lohse A, Rostamzadeh A, Metzger C, Munk MH, Peters O, Preis L, Priller J, Scheffler K, Schneider A, Spottke A, Spruth EJ, Ramirez A, Roske S, Roy N, Teipel S, Wagner M, Wiltfang J, Wolfsgruber S, Yakupov R, Zeidman P, Jessen F, Schott BH, Duzel E, Maass A; DELCODE Study Group. Novelty-Related fMRI Responses of Precuneus and Medial Temporal Regions in Individuals at Risk for Alzheimer Disease. Neurology. 2022 Aug 23;99(8):e775-e788. doi: 10.1212/WNL.0000000000200667. Epub 2022 Jun 3. PMID 35995589
- [Background] Buzsaki G, Wang XJ. Mechanisms of gamma oscillations. Annu Rev Neurosci. 2012;35:203-25. doi: 10.1146/annurev-neuro-062111-150444. Epub 2012 Mar 20. PMID 22443509
- [Background] Celone KA, Calhoun VD, Dickerson BC, Atri A, Chua EF, Miller SL, DePeau K, Rentz DM, Selkoe DJ, Blacker D, Albert MS, Sperling RA. Alterations in memory networks in mild cognitive impairment and Alzheimer's disease: an independent component analysis. J Neurosci. 2006 Oct 4;26(40):10222-31. doi: 10.1523/JNEUROSCI.2250-06.2006. PMID 17021177
- [Background] Damoiseaux JS, Beckmann CF, Arigita EJ, Barkhof F, Scheltens P, Stam CJ, Smith SM, Rombouts SA. Reduced resting-state brain activity in the "default network" in normal aging. Cereb Cortex. 2008 Aug;18(8):1856-64. doi: 10.1093/cercor/bhm207. Epub 2007 Dec 5. PMID 18063564
- [Background] De Marco M, Ourselin S, Venneri A. Age and hippocampal volume predict distinct parts of default mode network activity. Sci Rep. 2019 Nov 5;9(1):16075. doi: 10.1038/s41598-019-52488-9. PMID 31690806
- [Background] Fell J, Klaver P, Lehnertz K, Grunwald T, Schaller C, Elger CE, Fernandez G. Human memory formation is accompanied by rhinal-hippocampal coupling and decoupling. Nat Neurosci. 2001 Dec;4(12):1259-64. doi: 10.1038/nn759. PMID 11694886
- [Background] Flanagin VL, Klinkowski S, Brodt S, Graetsch M, Roselli C, Glasauer S, Gais S. The precuneus as a central node in declarative memory retrieval. Cereb Cortex. 2023 May 9;33(10):5981-5990. doi: 10.1093/cercor/bhac476. PMID 36610736
- [Background] Gaetz W, Roberts TP, Singh KD, Muthukumaraswamy SD. Functional and structural correlates of the aging brain: relating visual cortex (V1) gamma band responses to age-related structural change. Hum Brain Mapp. 2012 Sep;33(9):2035-46. doi: 10.1002/hbm.21339. Epub 2011 Jul 18. PMID 21769992
- [Background] Gillespie AK, Jones EA, Lin YH, Karlsson MP, Kay K, Yoon SY, Tong LM, Nova P, Carr JS, Frank LM, Huang Y. Apolipoprotein E4 Causes Age-Dependent Disruption of Slow Gamma Oscillations during Hippocampal Sharp-Wave Ripples. Neuron. 2016 May 18;90(4):740-51. doi: 10.1016/j.neuron.2016.04.009. Epub 2016 May 5. PMID 27161522
- [Background] Griffiths BJ, Parish G, Roux F, Michelmann S, van der Plas M, Kolibius LD, Chelvarajah R, Rollings DT, Sawlani V, Hamer H, Gollwitzer S, Kreiselmeyer G, Staresina B, Wimber M, Hanslmayr S. Directional coupling of slow and fast hippocampal gamma with neocortical alpha/beta oscillations in human episodic memory. Proc Natl Acad Sci U S A. 2019 Oct 22;116(43):21834-21842. doi: 10.1073/pnas.1914180116. Epub 2019 Oct 9. PMID 31597741
- [Background] Hebscher M, Meltzer JA, Gilboa A. A causal role for the precuneus in network-wide theta and gamma oscillatory activity during complex memory retrieval. Elife. 2019 Feb 11;8:e43114. doi: 10.7554/eLife.43114. PMID 30741161
- [Background] Heusser AC, Poeppel D, Ezzyat Y, Davachi L. Episodic sequence memory is supported by a theta-gamma phase code. Nat Neurosci. 2016 Oct;19(10):1374-80. doi: 10.1038/nn.4374. Epub 2016 Aug 29. PMID 27571010
- [Background] Hijazi S, Smit AB, van Kesteren RE. Fast-spiking parvalbumin-positive interneurons in brain physiology and Alzheimer's disease. Mol Psychiatry. 2023 Dec;28(12):4954-4967. doi: 10.1038/s41380-023-02168-y. Epub 2023 Jul 7. PMID 37419975
- [Background] Hu H, Gan J, Jonas P. Interneurons. Fast-spiking, parvalbumin(+) GABAergic interneurons: from cellular design to microcircuit function. Science. 2014 Aug 1;345(6196):1255263. doi: 10.1126/science.1255263. Epub 2014 Jul 31. PMID 25082707
- [Background] Huang D, Liu D, Yin J, Qian T, Shrestha S, Ni H. Glutamate-glutamine and GABA in brain of normal aged and patients with cognitive impairment. Eur Radiol. 2017 Jul;27(7):2698-2705. doi: 10.1007/s00330-016-4669-8. Epub 2016 Dec 13. PMID 27966041
- [Background] Jimenez-Balado J, Ycaza Herrera A, Igwe K, Klem L, Buyukturkoglu K, Irimia A, Chen L, Guo J, Brickman AM, Eich TS. Reduced Hippocampal GABA+ Is Associated With Poorer Episodic Memory in Healthy Older Women: A Pilot Study. Front Behav Neurosci. 2021 Aug 26;15:695416. doi: 10.3389/fnbeh.2021.695416. eCollection 2021. PMID 34512283
- [Background] Kawaguchi Y, Katsumaru H, Kosaka T, Heizmann CW, Hama K. Fast spiking cells in rat hippocampus (CA1 region) contain the calcium-binding protein parvalbumin. Brain Res. 1987 Jul 28;416(2):369-74. doi: 10.1016/0006-8993(87)90921-8. PMID 3304536
- [Background] Kircher TT, Weis S, Freymann K, Erb M, Jessen F, Grodd W, Heun R, Leube DT. Hippocampal activation in patients with mild cognitive impairment is necessary for successful memory encoding. J Neurol Neurosurg Psychiatry. 2007 Aug;78(8):812-8. doi: 10.1136/jnnp.2006.104877. Epub 2007 Feb 7. PMID 17287238
- [Background] Klunk WE, Engler H, Nordberg A, Wang Y, Blomqvist G, Holt DP, Bergstrom M, Savitcheva I, Huang GF, Estrada S, Ausen B, Debnath ML, Barletta J, Price JC, Sandell J, Lopresti BJ, Wall A, Koivisto P, Antoni G, Mathis CA, Langstrom B. Imaging brain amyloid in Alzheimer's disease with Pittsburgh Compound-B. Ann Neurol. 2004 Mar;55(3):306-19. doi: 10.1002/ana.20009. PMID 14991808
- [Background] Lundstrom BN, Ingvar M, Petersson KM. The role of precuneus and left inferior frontal cortex during source memory episodic retrieval. Neuroimage. 2005 Oct 1;27(4):824-34. doi: 10.1016/j.neuroimage.2005.05.008. PMID 15982902
- [Background] Murty DVPS, Manikandan K, Kumar WS, Ramesh RG, Purokayastha S, Javali M, Rao NP, Ray S. Gamma oscillations weaken with age in healthy elderly in human EEG. Neuroimage. 2020 Jul 15;215:116826. doi: 10.1016/j.neuroimage.2020.116826. Epub 2020 Apr 7. PMID 32276055
- [Background] Nyberg L, Lovden M, Riklund K, Lindenberger U, Backman L. Memory aging and brain maintenance. Trends Cogn Sci. 2012 May;16(5):292-305. doi: 10.1016/j.tics.2012.04.005. PMID 22542563
- [Background] Oeltzschner G, Wijtenburg SA, Mikkelsen M, Edden RAE, Barker PB, Joo JH, Leoutsakos JS, Rowland LM, Workman CI, Smith GS. Neurometabolites and associations with cognitive deficits in mild cognitive impairment: a magnetic resonance spectroscopy study at 7 Tesla. Neurobiol Aging. 2019 Jan;73:211-218. doi: 10.1016/j.neurobiolaging.2018.09.027. Epub 2018 Sep 27. PMID 30390554
- [Background] Palop JJ, Mucke L. Network abnormalities and interneuron dysfunction in Alzheimer disease. Nat Rev Neurosci. 2016 Dec;17(12):777-792. doi: 10.1038/nrn.2016.141. Epub 2016 Nov 10. PMID 27829687
- [Background] Porges EC, Woods AJ, Edden RA, Puts NA, Harris AD, Chen H, Garcia AM, Seider TR, Lamb DG, Williamson JB, Cohen RA. Frontal Gamma-Aminobutyric Acid Concentrations Are Associated With Cognitive Performance in Older Adults. Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Jan;2(1):38-44. doi: 10.1016/j.bpsc.2016.06.004. PMID 28217759
- [Background] Riese F, Gietl A, Zolch N, Henning A, O'Gorman R, Kalin AM, Leh SE, Buck A, Warnock G, Edden RA, Luechinger R, Hock C, Kollias S, Michels L. Posterior cingulate gamma-aminobutyric acid and glutamate/glutamine are reduced in amnestic mild cognitive impairment and are unrelated to amyloid deposition and apolipoprotein E genotype. Neurobiol Aging. 2015 Jan;36(1):53-9. doi: 10.1016/j.neurobiolaging.2014.07.030. Epub 2014 Jul 29. PMID 25169676
- [Background] Sederberg PB, Schulze-Bonhage A, Madsen JR, Bromfield EB, McCarthy DC, Brandt A, Tully MS, Kahana MJ. Hippocampal and neocortical gamma oscillations predict memory formation in humans. Cereb Cortex. 2007 May;17(5):1190-6. doi: 10.1093/cercor/bhl030. Epub 2006 Jul 10. PMID 16831858
- [Background] Wagner AD, Shannon BJ, Kahn I, Buckner RL. Parietal lobe contributions to episodic memory retrieval. Trends Cogn Sci. 2005 Sep;9(9):445-53. doi: 10.1016/j.tics.2005.07.001. PMID 16054861